CLINICAL TRIAL: NCT02172924
Title: A Phase 2 Study Using Placenta Derived Decidual Stromal Cells for Graft Versus Host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Olle Ringdén, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSCGVHD001
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Graft vs Host Disease
Keywords: Stem Cell Transplantation; Decidual Stromal Cells
MeSH Terms: conditions — Graft vs Host Disease

ARMS (2):
- Early Decidual Stromal Cells (Active Comparator): Patients with therapy-refractory GVHD and on calcineurin inhibitor and high dose corticosteroids since no more than 7 days will be given Decidual Stromal Cell therapy.
  Interventions: Biological: Early Decidual stromal cell therapy
- Late Decidual Stromal Cells (Active Comparator): Patients with therapy-refractory GVHD and on calcineurin inhibitor and high dose corticosteroids for longer than 7 days will be given Decidual Stromal Cell therapy.
  Interventions: Biological: Late Decidual stromal cell therapy

INTERVENTIONS:
Biological: Early Decidual stromal cell therapy — Intervention given within 7 days after corticosteroids.
  Arms: Early Decidual Stromal Cells
Biological: Late Decidual stromal cell therapy — Intervention given after 7 days after corticosteroids.
  Arms: Late Decidual Stromal Cells

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy using decidual stromal cell therapy for graft versus host disease after allogeneic hematopoietic stem cell transplantation. The hypothesis to be tested is that the cells are safe to infuse and that they have a positive clinical effect.

DETAILED DESCRIPTION:
Patients with GVHD grade 2-4, will receive decidual stromal cells at approximately 1x10^6 cells/kg at one or more occasions at weekly intervals dependent on clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Acute graft versus host disease grade 2-4 or therapy resistant chronic graft versus host disease.
* Are on calcineurin inhibitor and high dose corticosteroids.

Exclusion Criteria:

* Terminally ill patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Actuarial survival at one year after onset of graft versus host disease | 12 months after inclusion

SECONDARY OUTCOMES:
Response at 28 days after onset of graft versus host disease | 28 days after inclusion
Side effects | Up to 6 months after inclusion
Incidence of severe infections | Up to 12 months after inclusion
Disease free survival | 12 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringdén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden